CLINICAL TRIAL: NCT05904951
Title: Balloon Dilatation Catheter for the Dilation of Stenotic Atherosclerotic Lesions in Coronary Artery or Bypass Grafts: Evaluation of Safety and Performance in Everyday Clinical Practice. The INVADER™ Percutaneous Transluminal Coronary Angioplasty (PTCA) Post Market Clinical Follow-up (PMCF) Study
Brief Title: The INVADER™ Percutaneous Transluminal Coronary Angioplasty (PTCA) Post Market Clinical Follow-up (PMCF) Study
Status: Completed | Type: Observational
Sponsor: Alvimedica (Industry)
Responsible Party: Sponsor
Other Study IDs: C32104
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Coronary Disease; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: INVADER™ PTCA Balloon Dilatation Catheter — INVADER™ PTCA Balloon Dilatation Catheter is a single use, EO sterilized, monorail rapid exchange (RX) coronary angioplasty balloon dilatation catheter. The INVADER™ PTCA has been designed to dilate the stenotic atherosclerotic lesions in coronary arteries or bypass grafts. The INVADER™ PTCA is an interventional, non-surgical device, and considered minimally invasive.

SUMMARY:
The aim of the present observational study is to collect clinical data on the non-implantable medical device INVADER™ PTCA in the daily use in an unselected population.

ELIGIBILITY:
Inclusion Criteria:

* To be a Turkish citizen,
* To be >18 years of age,
* Lesion must be successfully crossed with a guidewire without complication,
* INVADER™ PTCA is used in the primary lesion treated during the procedure,
* Patient has signed and dated the informed consent.

Exclusion Criteria:

* Patients who have a known allergic reaction to any of the composition of INVADER™ PTCA Balloon Dilatation Catheter.
* Device use not consistent with Instructions for Use (IFU).
* Patients concurrently participating in another medical device or pharmaceutical clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of all consecutive patients treated with the INVADER™ PTCA at the study sites: all patients who met the inclusion/exclusion criteria were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Device success | 48 hours after index procedure
  Measurement: Percentage of lesions among all attempted lesions with:
  * Successful device delivery, and
  * Successful inflation, achievement of appropriate diameter, and deflation of the balloon, and
  * Decrease in the percent stenosis after balloon procedure, and
  * No perforation, flow-limiting dissection or reduction in TIMI flow grade, and
  * No life-threatening arrhythmias (sustained ventricular tachycardia, ventricular fibrillation)

SECONDARY OUTCOMES:
Rate of individual components of device success | 48 hours after index procedure
Procedural success: | 48 hours after index procedure
  o Measurement: Percentage of device success without major adverse cardiovascular events (MACE) (composite of all death, myocardial infarction [MI], and clinically indicated target lesion revascularization [CI-TLR]).
Rate of Target Lesion Failure (TLF) | 48 hours after index procedure
  o Measurement: Percentage of a composite of cardiac death, target vessel myocardial infarction (TV-MI), and CI-TLR.

CONTACTS AND LOCATIONS:
Locations (1):
- Alvimedica, Istanbul, Turkey (Türkiye)